CLINICAL TRIAL: NCT06890936
Title: Clinical Characteristics and Outcomes of Patients Requiring Mechanical Ventilation- a Nepalese Single Center Retrospective Study of 5 Years.
Brief Title: Clinical Characteristics and Outcomes of Patients Requiring Mechanical Ventilation in an ICU- a Registry Based Study
Status: Completed | Type: Observational
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Bipin Karki, Dr., Tribhuvan University Teaching Hospital, Institute Of Medicine.
Other Study IDs: 397(6-11)E2-081/082
Record Dates: First submitted 2025-03-16; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Mechanical Ventilation; Intensive Care Unit
Keywords: mechanical ventilation; intensive care unit; outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MV: Patients requiring mechanical ventilation

SUMMARY:
Rationale: Patients admitted to the Intensive Care Unit (ICU) often require respiratory support in terms of mechanical ventilation (either non-invasive or invasive). Though these patients may be diverse in clinical characteristics, the need of respiratory support in itself is in many conditions a factor relating poorer outcomes. The exact association of the requirement of respiratory support in our patient population is missing in the current literature. This study will look at 5-year data of patients admitted to the ICUs of Tribhuvan University Teaching Hospital and try to characterize these patients according to their clinical profile. Further, this study will also help to generate data regarding the outcomes of such patients.

Study Objective: To characterize the patients requiring respiratory support in the ICUs of TUTH and find their outcomes in terms of ICU mortality.

Design: A registry based, retrospective, descriptive, cohort study. Sample size: Convenience sampling of all the patients who are admitted to the ICU.

Duration: Retrospective data from the 5-year period between November 1, 2019 to December 31, 2024.

Place: Intensive care units (ICUs), Tribhuvan University Teaching Hospital (TUTH).

Interventions: Not applicable Expected results: The study will help determine the clinical characteristics of patients admitted to the ICUs of TUTH requiring respiratory support and their associated outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Admission to the ICU

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the ICU
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
ICU mortality | At the end of 5 years
  Mortality during ICU stay

CONTACTS AND LOCATIONS:
Locations (1):
- Tribhuvan University Teaching Hospital, Mahārājgañj, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Undecided